CLINICAL TRIAL: NCT00782470
Title: A Prospective, Non-interventional, Multi-center, Open-label Study to Evaluate the Reasons and Consequences of Bleeding in Late Teens and Early Adulthood Subjects With Severe Hemophilia A Receiving Prophylaxis and On-demand Treatment Regimen
Brief Title: Evaluation of the Reasons and Consequences of Bleeding in Late Teens and Early Adulthood Patients With Severe Hemophilia A
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 12749
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Hematologic Disease; Blood Coagulation Disorders
MeSH Terms: conditions — Hematologic Diseases; Blood Coagulation Disorders | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1
  Interventions: Behavioral: Recombinant Factor VIII (Kogenate, BAY 14-2222)
- Group 2
  Interventions: Behavioral: Recombinant Factor VIII (Kogenate, BAY 14-2222)
- Group 3
  Interventions: Behavioral: Recombinant Factor VIII (Kogenate, BAY 14-2222)

INTERVENTIONS:
Behavioral: Recombinant Factor VIII (Kogenate, BAY 14-2222) — Subjects electing to stay on the prophylactic treatment (prospective)
  Groups: Group 1
Behavioral: Recombinant Factor VIII (Kogenate, BAY 14-2222) — Subjects electing to switch to on-demand treatment (prospective)
  Groups: Group 2
Behavioral: Recombinant Factor VIII (Kogenate, BAY 14-2222) — Subjects remaining on-demand treatment (retrospective)
  Groups: Group 3

SUMMARY:
Understanding how often the bleeding events occur in the subjects who voluntarily decide to switch from prophylaxis to on-demand and in those subjects who remain on prophylaxis. Also look into the consequences of switching treatment in QoL (quality of life), development of target joints, activity level and reasons that might influence the desire to switch.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (<2%)
* For subjects who elect staying on Prophylaxis only: Have been on continuous prophylactic treatment for the past 5 years prior to study entry
* For subjects who elect switching to on-demand only: Have been on continuous prophylactic treatment for the past 5 years, but may have been on intermediate or reduced prophylaxis for the 1-12 months prior to study entry
* For subjects currently on-demand: a retrospective arm of subjects who have been on continuous prophylactic treatment for at least 5 years and switched to on-demand treatment between 13 and 24 months prior to study entry
* Current treatment with rFVIII

Exclusion Criteria:

* Other known hematological / bleeding disorders other than hemophilia A
* Participating on another study that may have an impact on bleeding or the objectives of this study
* Known alcohol and drug abuse

Ages: 14 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cohort 1 - Prospective Prophylaxis Group Cohort 2 - Prospective On-demand Group Cohort 3 - Retrospective On-demand Group
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the frequency of all bleeds (spontaneous and trauma) during the study | End of Study

SECONDARY OUTCOMES:
To evaluate the change from baseline in HRQoL (health-related quality of life) | End of Study
To evaluate number of patients that want to return to prophylaxis treatment after having switched to on-demand therapy | End of Study
To evaluate the change from baseline in the Gilbert score | End of Study
To evaluate the number of target joint development | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- United States (7):
  - Duarte, California
  - Denver, Colorado
  - Peoria, Illinois
  - Jefferson City, Missouri
  - Las Vegas, Nevada
  - Fort Worth, Texas
  - Houston, Texas
- Many Locations, Canada
- Many Locations, Germany
- Many Locations, United Kingdom

REFERENCES:
- [Result] Manco-Johnson MJ, Sanders J, Ewing N, Rodriguez N, Tarantino M, Humphries T; TEEN/TWEN Study Group. Consequences of switching from prophylactic treatment to on-demand treatment in late teens and early adults with severe haemophilia A: the TEEN/TWEN study. Haemophilia. 2013 Sep;19(5):727-35. doi: 10.1111/hae.12177. Epub 2013 Jun 11. PMID 23750875